CLINICAL TRIAL: NCT04743011
Title: Nebulized Enriched Heparin to Treat no Critical Patients With Sars-Cov-2 - Triple Blind Clinical Trial
Brief Title: Enriched Heparin Anti COVID-19 Trial
Acronym: EnHanCed
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Principal Investigator, Matheus Bertanha, PhD, Principal Investigator, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPECLIN-MB-2
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Covid19
Keywords: COVID-19; Heparin; Antiviral Agents; Blood Coagulation; Clinical Protocols
MeSH Terms: conditions — COVID-19; Thrombosis | interventions — Heparin; Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants allocated to Group 1 (control) will receive inhalation with 0.9% saline solution applied 4/4 hours, for 7 days. Participants allocated to Group 2 (intervention) will receive high molecular weight inhaled heparin (2,5mg / mL 0.9% SF), at a 4/4 hour dose, for 7 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The clinical trial will be triple-blind. Participants, researchers, and the data/statistical analysis team will not have access to the research data. Only one member of the team will produce the test product and assist a external physician (not part of the research team), with the adverse events that may occur with the participants during the execution of the research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive inhalation with 5mL 0.9% saline solution (placebo), 4/4h, during the day period (5 doses).
  Interventions: Drug: Placebo
- Heparin sodium (Active Comparator): Participants will receive inhalation with 5mL 0.9% saline solution + 2,5mg of high molecular weight heparin - enriched heparin, 4/4h, during the day period (5 doses).
  Interventions: Drug: Heparin sodium

INTERVENTIONS:
Drug: Heparin sodium — Nebulized inhalation of 5 mL of a solution containing high molecular weight heparin - enriched heparin - 2.5mg/mL and 0.9% saline solution, every 4 hours for 7 days, except during the nighttime (5 doses/day)
  Other Names: Hepamax S BLAU
  Arms: Heparin sodium
Drug: Placebo — Nebulized inhalation of 5 mL of 0.9% saline solution, every 4 hours for 7 days, except during the nighttime (5 doses/day)
  Other Names: Saline solution 0.9%; Physiological solution 0.9%
  Arms: Placebo

SUMMARY:
Coronavirus 19 (COVID-19) is a viral respiratory disease that was identified in December 2019 after the first cases in China, spreading rapidly until reaching pandemic status, causing the collapse of numerous health systems and strong economic and social impact. By the end of April 2020, 3.08 million cases, and more than 214 thousand deaths were already recorded. The treatment so far has not been established and there are several clinical trials testing known drugs that have antiviral activity in vitro, due to the urgency that the global situation imposes. Medicines with specific actions can take years to be discovered, while a vaccine also takes a long time. Recently, it has been shown that the worsening of Coronavirus infection may be related to the formation of micro clots in blood vessels and anticoagulants have been used as adjuvants in the treatment. This study is justified by conducting a pilot study that showed an in vitro antiviral action (anti-COVID-19) of high molecular weight heparin. Methods: A phase I / II clinical trial will be conducted. 40 participants will be included in two arms. Participants allocated to Group 1 (control) will receive inhalation with 0.9% saline applied 4/4 hours, for 7 days. Participants allocated to Group 2 (intervention) will receive high molecular weight inhaled heparin (250ug / mL 0.9% SF), at a 4/4 hour dose, for 7 days. The outcomes of interest will be safety (absence of moderate or serious adverse events) and effectiveness (measured in a score of 7 points, with 1 absence of limitations and 7, death). Expected results: The development of a new therapeutic option for COVID-19 is expected, with the possibility of use in other serious coronavirus diseases, to be subsequently tested in phase III studies.

DETAILED DESCRIPTION:
In view of the enormous health, financial and social crisis resulting of the pandemic caused by SARS-Cov-2, it is justified to urgently conduct tests with possible antiviral drugs. The high molecular weight heparin (HMWH) (heparin enriched by ultrafiltration process) proposed by this study, has a potential inhibition activity over viral replication, demonstrated by preliminary in vitro tests, carried out in a model established in partnership with the Laboratory of Clinical and Molecular Virology (LVCM) of the Institute of Biomedical Sciences of the University of São Paulo (ICB-USP).

Along with the findings in the literature, such as the study carried out by Phelps, M.K. et al (2020), among others, the use of inhaled heparin presents adequate levels of safety to be used in a clinical trial. Taking into account that the dose of high molecular weight heparin (enriched by this study team) with antiviral activity in vitro is much lower than the doses currently presented in published clinical trials using inhaled UFH, we have the safety premise to carry out this study. The intentions of this study differ from what has been presented in the world literature so far, as it does not aim to induce anticoagulation, nor to effectively inhibit the formation of pulmonary fibrin, but rather, to act as an inhibitor of viral replication.

Also, as characteristics of the product to be tested, this heparin (HMWH) is presented in a buffered solution free of low-sulfated low-weight molecules, which is obtained in a sterile environment through ultrafiltration of the unfractionated solution of porcine origin available in Brazil (Hemofol - Cristália) using Centriprep-10kDa® centrifuge filter (Millipore ™) used as recommended by the manufacturer.

The high molecular weight heparin (HMWH) - enriched heparin - had two process patents filed, one under the description "HIGH MOLECULAR WEIGHT DEFINITION HEPARINE DEVELOPMENT PROCESS", BR 102014027804-4 A2 - granted by the Instituto Nacional de Propriedade Industrial (INPI) and another with the description "COMPOSITION OF HIGH MOLECULAR WEIGHT NON-FRACTIONAL HEPARINE FOR ANTIVIRAL ACTION ", BR 102020 011964-8 - deposited at INPI.

ELIGIBILITY:
Inclusion Criteria:

* Signature and agreement to the Free Consent Form;
* Both sexes, of any ethnic origin, aged between 18 and 90 years;
* COVID-19 infected patients diagnosed by RT-PCR (reverse-transcriptase polymerase chain reaction) or with a strong suspicion of COVID-19 by clinical evaluation through compatible clinical and radiological findings;
* Time of disease evolution less than 10 days;
* Radiological diagnosis of grade 2A pneumonia, with gas exchange ratio > 200 on blood gas analysis (paO2 / pFiO2), characterizing mild hypoxemia;
* Indication of hospital treatment regime, provided that the period of hospitalization before inclusion is not more than 24 hours;
* Need for supplemental oxygen therapy (O2) less than 5L / min.

Exclusion Criteria:

* No agreement to the terms of this study;
* Moderate or severe respiratory failure requiring admission to the ICU and the need for invasive mechanical ventilation or non-invasive ventilation (NIV) with positive pressure;
* Pregnancy or puerperium;
* Patients with hematological diseases, coagulation disorders, use of anticoagulants, previous heparin-induced allergy or thrombocytopenia, thrombocytopenia with a count of fewer than 50,000 platelets / mm3;
* COVID-19 not confirmed by RT-PCR within 72 hours of inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matheus Bertanha, PhD, Principal Investigator — São Paulo State University (Unesp)
Locations (2):
- Brazil (2):
  - School of Medicine at Botucatu- Paulista State University- UNESP, São Paulo, Brazil, Botucatu, São Paulo
  - Hospital das Clinicas de Boucatu, Botucatu, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The summary data will be published or made available 6 months after publication.
Access Criteria: Epidemiological data, clinical data, and patient evolution will be shared during the study only for researchers who request access to the data. Access requests will be analyzed by the main researcher, and they will only be released for scientific purposes.

REFERENCES:
- [Background] Phelps MK, Olson LM, Patel MAVB, Thompson MJ, Murphy CV. Nebulized Heparin for Adult Patients With Smoke Inhalation Injury: A Review of the Literature. J Pharm Technol. 2020 Aug;36(4):130-140. doi: 10.1177/8755122520925774. Epub 2020 Jun 1. PMID 34752548
- [Derived] Ramos da Silva Grillo VT, Bertanha M, da Silva Rodrigues L, de Lima MA, Mellucci Filho PL, Rahal Guaragna Machado R, Durigon EL, Dias Sertorio N, de Assis Golim M, Moroz A, Marques Braz AM, de Moraes LN, Leite MA, Bonciani Nader H, de Campos GC, Rodrigues Guzzo Carvalho C, Florenca Cardoso F, Magro AJ, Caputo Nunes H, Tommasini Grotto RM, de Cassia Alvarado R, de Moura Campos Pardini MI, Lima Sobreira M, da Costa EAPN, Naime Barbosa A, Fortaleza CMCB. Nebulized enriched heparin improves respiratory parameters in patients with COVID-19: a phase I/II randomized and triple-blind clinical trial. Sci Rep. 2024 Aug 27;14(1):19902. doi: 10.1038/s41598-024-70064-8. PMID 39191809

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Heparin Sodium
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Heparin Sodium | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Full Range); unit: years] | 52 [33 to 79] | 53 [27 to 84] | 53 [27 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 8 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 13 | 25
  Black | 2 | 0 | 2
Weight [Mean (Full Range); unit: kilograms] | 92 [67 to 132] | 79 [40 to 120] | 85 [40 to 132]
Height [Mean (Full Range); unit: centimeters] | 168 [150 to 183] | 162 [138 to 177] | 165 [138 to 183]
Body Mass Index [Mean (Full Range); unit: kg/m²] | 33 [24.3 to 52.9] | 29.4 [18.2 to 44.1] | 31.3 [18.2 to 52.9]
Hypertension [Count of Participants; unit: Participants] | 10 | 5 | 15
Coronary Disease [Count of Participants; unit: Participants] | 3 | 1 | 4
Dyslipidemia [Count of Participants; unit: Participants] | 6 | 9 | 15
Sedentarism [Count of Participants; unit: Participants] | 12 | 10 | 22
Tabagism [Count of Participants; unit: Participants] | 2 | 1 | 3
Previous Tabagism (Ceased) [Count of Participants; unit: Participants] | 2 | 4 | 6
Alcoholism [Count of Participants; unit: Participants] | 0 | 2 | 2
Previous Stroke [Count of Participants; unit: Participants] | 1 | 1 | 2
Previous Cancer [Count of Participants; unit: Participants] | 0 | 0 | 0
Previous Transplantation or Immunosuppression [Count of Participants; unit: Participants] | 3 | 3 | 6
Autoimmune Disease [Count of Participants; unit: Participants] | 0 | 1 | 1
Pulmonary Emphysema or Asthma [Count of Participants; unit: Participants] | 2 | 1 | 3
Hypothyroidism [Count of Participants; unit: Participants] | 0 | 2 | 2
Anxiety or Depression Disorders [Count of Participants; unit: Participants] | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Activated Partial Thromboplastin Time (APTT) > 1.5 Seconds
Description: Safety-related to the use of high molecular weight heparin inhaled in patients with SARS-COV-2 through the assessment of hemorrhagic events of any nature, alteration of the coagulogram that indicates an APTT ratio > 1.5 or heparin-induced thrombocytopenia.
  In Brazilian standards, the APTT is measured in seconds and compared to a laboratory control for a ratio, which is used as a measurement.
Time Frame: Immediately or up to 8 days after starting treatment
Measure: Mean (Full Range); unit: ratio
Arm/Group | Placebo | Heparin Sodium
Number analyzed (Participants) | 14 | 13
ratio | 0.95 [0.74 to 1.37] | 1.10 [0.88 to 1.45]

2. Primary Outcome: Number of Participants With a Negative Viral Load in Nasal Swab Reverse Transcription Polymerase Chain Reaction (RT-PCR).
Description: Effectiveness related to the proposed treatment, based on the analysis of the viral load of SARS-COV-2 virus in the participants through a sequential assessment of the viral load in nasal swab RT-PCR.
  The measurement consists in patients that tested negative for any viral load at the end of the treatment.
Time Frame: Immediately or up to 8 days after starting treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Heparin Sodium
Number analyzed (Participants) | 14 | 13
Participants | 8 | 8

3. Secondary Outcome: Number of Participants That Develop Renal Failure
Description: Worsening of clinical parameters characterized by renal failure through measurement of urea and creatinine;
Time Frame: Immediately or up to 8 days after starting treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Heparin Sodium
Number analyzed (Participants) | 14 | 13
Participants | 0 | 0

4. Secondary Outcome: Number of Participants That Develop Major Cardiovascular Events
Description: Worsening of clinical parameters characterized by major cardiovascular events (pulmonary embolism, acute myocardial infarction)
Time Frame: Immediately or up to 8 days after starting treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Heparin Sodium
Number analyzed (Participants) | 14 | 13
Participants | 0 | 0

5. Secondary Outcome: Number of Participants That Develop Deep Vein Thrombosis (DVT)
Description: Worsening of clinical parameters characterized by deep vein thrombosis (DVT);
Time Frame: Immediately or up to 8 days after starting treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Heparin Sodium
Number analyzed (Participants) | 14 | 13
Participants | 0 | 0

6. Secondary Outcome: Number of Participants That Develop Pancreatitis
Description: Worsening of clinical parameters characterized by pancreatitis through measurement of amylase (> 200 U/L);
Time Frame: Immediately or up to 8 days after starting treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Heparin Sodium
Number analyzed (Participants) | 14 | 13
Participants | 0 | 0

7. Secondary Outcome: Number of Deaths Among Participants
Description: Worsening of clinical parameters characterized by death;
Time Frame: Immediately or up to 8 days after starting treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Heparin Sodium
Number analyzed (Participants) | 14 | 13
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Increased C Reactive Protein Test
Description: Worsening of laboratory parameters measured by increase in C reactive protein test (>3.00mg/L);
Time Frame: Immediately or up to 8 days after starting treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Heparin Sodium
Number analyzed (Participants) | 14 | 13
Participants | 2 | 2

9. Secondary Outcome: Number of Participants With Deterioration of Arterial Blood Gas paO2/pFiO2 Ratio
Description: Worsening of laboratory parameters measured by alterations in arterial blood gas measured by paO2/pFiO2 < 200;
Time Frame: Immediately or up to 8 days after starting treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Heparin Sodium
Number analyzed (Participants) | 14 | 13
Participants | 1 | 1

10. Secondary Outcome: Number of Participants With Increased Pulmonary Area Compromised (%)
Description: Worsening of tomographic parameters measured by the pulmonary area compromised by the infection and/or inflammation.
Time Frame: Immediately or up to 8 days after starting treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Heparin Sodium
Number analyzed (Participants) | 14 | 13
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: No adverse effects were reported during the time frame of 7 days in which the groups were monitored.
Arm/Group | Placebo | Heparin Sodium
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT04743011/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT04743011/ICF_001.pdf